CLINICAL TRIAL: NCT06346119
Title: Evaluation of the Impact of Touch Relaxation in Sedated Intubated Patients Hospitalized in Intensive Care at Niort Hospital
Acronym: ETDR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Niort (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PI-2023-01
Record Dates: First submitted 2023-01-05; First posted 2024-04-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Reaction Anxiety; Difficult or Failed Intubation
Keywords: chemical restraint; intensive care; intubation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study will be conducted in two parallel groups. At the inclusion, each patient will be assigned to one of two groups by randomization; one group will receive the "touch" and the second group will not receive it will be the control arm.
Who Masked: Outcomes Assessor
Masking Description: It's a person external to the care service and to the randomization process will collect the possible prescription of a chemical restraint or the evolution of this chemical restraint by the resuscitator, in order to maintain the blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): this arm will not received relaxing touch. It's a control arm
- Experimental (Experimental): this arm will received relaxing touch twice a day
  Interventions: Other: this arm will received relaxing touch (hands, feet, head) during 30 minutes twice a day

INTERVENTIONS:
Other: this arm will received relaxing touch (hands, feet, head) during 30 minutes twice a day — Patients who will be included in this arm will receive massage twice a day of the head (10 minutes), feet (10 minutes) and hands (10 minutes)
  Arms: Experimental

SUMMARY:
This is a randomized prospective study. This objective is the impact of "relaxing touch" on the use of chemical restraint for patients in intensive care from the lifting of sedation until extubation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age
* Intubated and sedated man or woman
* Extubation within 48 hours
* Intubation of more than 48 hours in total
* Patient in intensive care at Niort hospital
* The trusted person or referent accepting the patient's participation
* Patient affiliated to the social security system

Exclusion Criteria:

* Known pregnancy
* Patient who refused to participate in the study after the fact
* Patients under long-term antidepressant treatment (treatment longer than 3 months)
* Patients under guardianship or curatorship
* Patient deprived of liberty
* Skin lesions on the hands/feet/head (wounds, erythema, burns, bedsores, phlyctenes)
* Inclusion in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
chemical restraint | 1 year
  Comparison of the proportion of patients who received chemical restraint during the sedation release phase until extubation between the two groups (experimental and control arms)

SECONDARY OUTCOMES:
self-extubations | 1 year
  Comparison of the proportion of self-extubations between the 2 groups
patient discomfort | T=0, T=30 nimutes, T=60 minutes, T= 90 minutes
  Comparison of patient discomfort parameters between the 2 groups. The discomfort will be evaluated thank to body expression (unrest) and facial expression according to the BPS scale. The BPS scale is a behavioral pain scale used in intensive care for the sedated and ventilated adult patient.
  There discomfort parameters will be evaluated immediately after the relaxation touch, 30 min after, 60 min after and 90 min after.
  The patients included in a experimal group will be relaxation touch twice per day 12 hours apart
respiratory rate | T=0, T=30 nimutes, T=60 minutes, T= 90 minutes
  Comparison of vital parameters between the 2 groups. Comparison between respiratory rate (/min), cardiac rate (/min), pressur (mmHG), and ventilation mode.
  Touch could relax patients and thus lower the values of vital parameters. The patients included in a experimal group will be relaxation touch twice per day 12 hours apart
Ratio chemical restraint use | 1 year
  Ratio per patient corresponding to the number of days with chemical restraint use between inclusion and exclusion/total number of days between inclusion and extubation.
cardiac frequency | T=0, T=30 nimutes, T=60 minutes, T= 90 minutes
  Comparison of vital parameters between the 2 groups. Comparison between respiratory rate (/min), cardiac rate (/min), pressur (mmHG), and ventilation mode.
  Touch could relax patients and thus lower the values of vital parameters. The patients included in a experimal group will be relaxation touch twice per day 12 hours apart

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc M. Le Guevel, Nurse coordinator, Principal Investigator — Centre Hospitalier de Niort - France
Locations (1):
- Centre Hospitalier de Niort, Niort, France

IPD SHARING:
Plan to Share IPD: No